CLINICAL TRIAL: NCT02032030
Title: SATISFY-SOS: Systematic Assessment and Targeted Improvement of Services Following Yearlong Surgical Outcomes Surveys
Brief Title: Systematic Assessment and Targeted Improvement of Services Following Yearlong Surgical Outcomes Surveys
Acronym: SATISFY-SOS
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael Avidan, Director, Institute of Quality Improvement, Research & Informatics (INQUIRI), Washington University School of Medicine
Other Study IDs: 201203088
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-06

CONDITIONS: Heart Attack; Cardiac Arrest; Congestive Heart Failure; Atrial Fibrillation; Angina; Deep Vein Thrombosis; Pulmonary Embolism; Respiratory Arrest; Respiratory Failure; Pneumonia; Gastrointestinal Bleed; Stomach Ulcer; Delirium; Stroke; Nerve Injury; Surgical Wound Infection
Keywords: quality of Life; pain; nausea; falls; intraoperative awareness; anesthesia awareness; cognition; activities of daily living; major morbidity; all-cause mortality
MeSH Terms: conditions — Myocardial Infarction; Heart Arrest; Heart Failure; Atrial Fibrillation; Angina Pectoris; Venous Thrombosis; Pulmonary Embolism; Apnea; Respiratory Insufficiency; Pneumonia; Gastrointestinal Hemorrhage; Stomach Ulcer; Delirium; Stroke; Surgical Wound Infection; Pain; Nausea; Intraoperative Awareness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Based on limited published epidemiological data, up to an alarming 1 in 50 surgical inpatients die within 30 postoperative days. Based on our own data from the B-Unaware (NCT00281489) and BAG-RECALL (NCT00682825) clinical trials, 30-day postoperative mortality among high-risk surgical patients is comparable to this at Barnes-Jewish Hospital, and 1-year mortality among high-risk surgical patients may be as high as 10%. Short- and intermediate-term postoperative mortality is therefore a pressing public health concern. Similarly, postoperative major morbidity - including delirium, stroke, myocardial infarction, atrial fibrillation, blood clots, renal dysfunction, wound infection, pneumonia, respiratory failure, loss of functionality, and chronic pain - occurs commonly and affects a substantial proportion of surgical patients, critically ill patients and patients undergoing procedures for chronic pain. Many factors associate strongly and independently with postoperative mortality and major morbidity: patient age, functional status, comorbid medical conditions, and duration and invasiveness of surgery, among others. It is a strategic priority to identify pre- and intraoperative risk factors that are subject to modification.

DETAILED DESCRIPTION:
The overarching purpose of SATISFY-SOS is to implement a rigorous process to assess short-term and intermediate-term outcomes of surgical and procedural patients who receive anesthesia services at Barnes-Jewish Hospital facilities, located in St. Louis, Missouri. Specifically, patients will be followed for major morbidity events, for mortality, and for quality of life up to a year following their procedures. Patients receiving anesthesia services will provide informed consent to participate in SATISFY-SOS. Each patient will have the opportunity to respond to a baseline quality of life survey as well as to two comprehensive post-procedure surveys. These surveys are conducted by either email, mail or via a telephone interview at 30-90 days post-procedure and again at one year. The survey questions are primarily comprised of standardized, validated, non-proprietary survey tools covering the following topics: general health, mental health, emotional health, physical health, pain, falls, major morbidity, and cognition.

In addition to collecting patient-reported outcomes, comprehensive medical record information for each patient beginning with the preoperative assessment and spanning throughout the surgery or procedure, hospitalization period, time spent in intensive care and follow-up clinic visits is incorporated into the database. Additionally, mortality data including cause of death for all patients will be ascertained via the National Death Index and from information in hospital records. This allows for meaningful, comprehensive electronic data query capabilities. Under the umbrella of the SATISFY-SOS initiative, we intend to implement specific evidence-based and patient-centered quality improvement programs, and to ensure that they are effective when implemented in routine clinical care. Additionally, future IRB-approved research projects can utilize de-identified SATISFY-SOS data.

All electronic data are collected from existing clinical records. The primary SATISFY-SOS database is hosted on a firewall-secured, HIPAA-compliant server within the Department of Anesthesiology at Washington University School of Medicine and maintained and managed by the departmental IT team. Access to the SATISFY-SOS data is restricted from web access and limited to only the project Informaticist, Data Manager, and Director.

Regular internal auditing of the data are conducted for validity and completeness on a monthly basis. On an annual basis, the consent process is audited. The data entered early in the registry are compared with data entered subsequently. Sensitivity analyses are performed to determine whether data are missing at random. It is planned to compare the data obtained from patient-reported outcomes against a sample of data in the medical records and against data obtained from a sample of patients contacted again by telephone. A data dictionary for key data fields is currently being compiled. Standard operating procedures have been developed for registry operations, patient recruitment, data collection, data management and data analysis. No adverse events attributable to this activity are envisioned. Multiple outcomes are being tracked; no specific sample size has been calculated. Sensitivity analyses are planned for missing or unavailable data. No imputation is currently planned. The statistical analyses will depend on the variables and outcomes of interest. This registry is currently IRB-approved for total enrollment of 36,000 patients. This is subject to subsequent expansion, pending IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* Surgical and procedural patients who require anesthesia services

Exclusion Criteria:

* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are attempting to recruit all-comers visiting our preoperative assessment clinic, with current daily enrollment rates approaching 60%.
Sampling Method: Non-Probability Sample
Enrollment: 73952 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
quality of life | 1 year
functional health | 1 year
falls | 1 year
cognition | 1 year
emotional health | 1 year
mental health | 1 year
physical health | 1 year
pain | 1 year
intraoperative awareness | 30-90 days
all-cause mortality | 1 year
surgical wound infection | 1 year
nerve injury | 30-90 days
stroke | 1 year
delirium | 30-90days
Stomach Ulcer | 30-90 days
Gastrointestinal Bleed | 30-90 days
Pneumonia | 1 year
Respiratory Failure | 1 year
Respiratory Arrest | 1 year
Pulmonary Embolism | 1 year
Deep Vein Thrombosis | 1 year
Angina | 1 year
Atrial Fibrillation | 1 year
Congestive Heart Failure | 1 year
Cardiac Arrest | 1 year
Heart Attack | 1 year

OTHER OUTCOMES:
Return to Work | 1 year
  Return to work after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, FCASA, Principal Investigator — Washington University School of Medicine; Anshuman Sharma, MD, Study Director — Washington University School of Medicine; Daniel Helsten, MD, Study Director — Washington University School of Medicine; Arbi Ben Abdallah, PhD, Study Director — Washington University School of Medicine; Troy Wildes, MD, Study Director — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Kertai MD, Pal N, Palanca BJ, Lin N, Searleman SA, Zhang L, Burnside BA, Finkel KJ, Avidan MS; B-Unaware Study Group. Association of perioperative risk factors and cumulative duration of low bispectral index with intermediate-term mortality after cardiac surgery in the B-Unaware Trial. Anesthesiology. 2010 May;112(5):1116-27. doi: 10.1097/ALN.0b013e3181d5e0a3. PMID 20418692
- [Background] Kertai MD, Palanca BJ, Pal N, Burnside BA, Zhang L, Sadiq F, Finkel KJ, Avidan MS; B-Unaware Study Group. Bispectral index monitoring, duration of bispectral index below 45, patient risk factors, and intermediate-term mortality after noncardiac surgery in the B-Unaware Trial. Anesthesiology. 2011 Mar;114(3):545-56. doi: 10.1097/ALN.0b013e31820c2b57. PMID 21293252
- [Background] Noordzij PG, Poldermans D, Schouten O, Bax JJ, Schreiner FA, Boersma E. Postoperative mortality in The Netherlands: a population-based analysis of surgery-specific risk in adults. Anesthesiology. 2010 May;112(5):1105-15. doi: 10.1097/ALN.0b013e3181d5f95c. PMID 20418691
- [Background] Guijarro R, Montes J, San Roman C, Arcelus JI, Barillari G, Granero X, Monreal M. Venous thromboembolism and bleeding after total knee and hip arthroplasty. Findings from the Spanish National Discharge Database. Thromb Haemost. 2011 Apr;105(4):610-5. doi: 10.1160/TH10-10-0645. Epub 2010 Dec 21. PMID 21174008
- [Background] Jafari SM, Huang R, Joshi A, Parvizi J, Hozack WJ. Renal impairment following total joint arthroplasty: who is at risk? J Arthroplasty. 2010 Sep;25(6 Suppl):49-53, 53.e1-2. doi: 10.1016/j.arth.2010.04.008. Epub 2010 May 31. PMID 20570102
- [Background] Mantilla CB, Horlocker TT, Schroeder DR, Berry DJ, Brown DL. Frequency of myocardial infarction, pulmonary embolism, deep venous thrombosis, and death following primary hip or knee arthroplasty. Anesthesiology. 2002 May;96(5):1140-6. doi: 10.1097/00000542-200205000-00017. PMID 11981154
- [Background] Parvizi J, Mui A, Purtill JJ, Sharkey PF, Hozack WJ, Rothman RH. Total joint arthroplasty: When do fatal or near-fatal complications occur? J Bone Joint Surg Am. 2007 Jan;89(1):27-32. doi: 10.2106/JBJS.E.01443. PMID 17200306
- [Background] Singh JA, Jensen MR, Harmsen WS, Gabriel SE, Lewallen DG. Cardiac and thromboembolic complications and mortality in patients undergoing total hip and total knee arthroplasty. Ann Rheum Dis. 2011 Dec;70(12):2082-8. doi: 10.1136/ard.2010.148726. Epub 2011 Oct 21. PMID 22021865
- [Background] Sabate S, Mases A, Guilera N, Canet J, Castillo J, Orrego C, Sabate A, Fita G, Parramon F, Paniagua P, Rodriguez A, Sabate M; ANESCARDIOCAT Group. Incidence and predictors of major perioperative adverse cardiac and cerebrovascular events in non-cardiac surgery. Br J Anaesth. 2011 Dec;107(6):879-90. doi: 10.1093/bja/aer268. Epub 2011 Sep 2. PMID 21890661
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Kheterpal S, Tremper KK, Heung M, Rosenberg AL, Englesbe M, Shanks AM, Campbell DA Jr. Development and validation of an acute kidney injury risk index for patients undergoing general surgery: results from a national data set. Anesthesiology. 2009 Mar;110(3):505-15. doi: 10.1097/ALN.0b013e3181979440. PMID 19212261
- [Background] Pearse RM, Holt PJ, Grocott MP. Managing perioperative risk in patients undergoing elective non-cardiac surgery. BMJ. 2011 Oct 5;343:d5759. doi: 10.1136/bmj.d5759. No abstract available. PMID 21976704
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Background] Brice DD, Hetherington RR, Utting JE. A simple study of awareness and dreaming during anaesthesia. Br J Anaesth. 1970 Jun;42(6):535-42. doi: 10.1093/bja/42.6.535. No abstract available. PMID 5423844
- [Background] Galvin JE, Roe CM, Powlishta KK, Coats MA, Muich SJ, Grant E, Miller JP, Storandt M, Morris JC. The AD8: a brief informant interview to detect dementia. Neurology. 2005 Aug 23;65(4):559-64. doi: 10.1212/01.wnl.0000172958.95282.2a. PMID 16116116
- [Background] Bruce J, Russell EM, Mollison J, Krukowski ZH. The measurement and monitoring of surgical adverse events. Health Technol Assess. 2001;5(22):1-194. doi: 10.3310/hta5220. PMID 11532239
- [Background] Gibbons C, Bruce J, Carpenter J, Wilson AP, Wilson J, Pearson A, Lamping DL, Krukowski ZH, Reeves BC. Identification of risk factors by systematic review and development of risk-adjusted models for surgical site infection. Health Technol Assess. 2011 Sep;15(30):1-156, iii-iv. doi: 10.3310/hta15300. PMID 21884656
- [Background] Best WR, Khuri SF, Phelan M, Hur K, Henderson WG, Demakis JG, Daley J. Identifying patient preoperative risk factors and postoperative adverse events in administrative databases: results from the Department of Veterans Affairs National Surgical Quality Improvement Program. J Am Coll Surg. 2002 Mar;194(3):257-66. doi: 10.1016/s1072-7515(01)01183-8. PMID 11893128
- [Background] Cima RR, Lackore KA, Nehring SA, Cassivi SD, Donohue JH, Deschamps C, Vansuch M, Naessens JM. How best to measure surgical quality? Comparison of the Agency for Healthcare Research and Quality Patient Safety Indicators (AHRQ-PSI) and the American College of Surgeons National Surgical Quality Improvement Program (ACS-NSQIP) postoperative adverse events at a single institution. Surgery. 2011 Nov;150(5):943-9. doi: 10.1016/j.surg.2011.06.020. Epub 2011 Aug 27. PMID 21875734
- [Background] Mashour GA, Shanks AM, Kheterpal S. Perioperative stroke and associated mortality after noncardiac, nonneurologic surgery. Anesthesiology. 2011 Jun;114(6):1289-96. doi: 10.1097/ALN.0b013e318216e7f4. PMID 21478735
- [Background] Mendis S, Thygesen K, Kuulasmaa K, Giampaoli S, Mahonen M, Ngu Blackett K, Lisheng L; Writing group on behalf of the participating experts of the WHO consultation for revision of WHO definition of myocardial infarction. World Health Organization definition of myocardial infarction: 2008-09 revision. Int J Epidemiol. 2011 Feb;40(1):139-46. doi: 10.1093/ije/dyq165. Epub 2010 Oct 5. PMID 20926369
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Bellomo R, Kellum JA, Ronco C. Defining and classifying acute renal failure: from advocacy to consensus and validation of the RIFLE criteria. Intensive Care Med. 2007 Mar;33(3):409-13. doi: 10.1007/s00134-006-0478-x. Epub 2006 Dec 13. PMID 17165018
- [Background] FLETCHER CM. Definition and classification of the causes of respiratory failure. Proc R Soc Med. 1962 Jul;55:565-6. No abstract available. PMID 13893562
- [Background] Gupta H, Gupta PK, Fang X, Miller WJ, Cemaj S, Forse RA, Morrow LE. Development and validation of a risk calculator predicting postoperative respiratory failure. Chest. 2011 Nov;140(5):1207-1215. doi: 10.1378/chest.11-0466. Epub 2011 Jul 14. PMID 21757571
- [Background] Consensus paper on the surveillance of surgical wound infections. The Society for Hospital Epidemiology of America; The Association for Practitioners in Infection Control; The Centers for Disease Control; The Surgical Infection Society. Infect Control Hosp Epidemiol. 1992 Oct;13(10):599-605. PMID 1334987
- [Derived] Fritz BA, Escallier KE, Ben Abdallah A, Oberhaus J, Becker J, Geczi K, McKinnon S, Helsten DL, Sharma A, Wildes TS, Avidan MS. Convergent Validity of Three Methods for Measuring Postoperative Complications. Anesthesiology. 2016 Jun;124(6):1265-76. doi: 10.1097/ALN.0000000000001108. PMID 27028469
- [Derived] Fritz BA, Kalarickal PL, Maybrier HR, Muench MR, Dearth D, Chen Y, Escallier KE, Ben Abdallah A, Lin N, Avidan MS. Intraoperative Electroencephalogram Suppression Predicts Postoperative Delirium. Anesth Analg. 2016 Jan;122(1):234-42. doi: 10.1213/ANE.0000000000000989. PMID 26418126